CLINICAL TRIAL: NCT06782971
Title: COSMOS-Avatar: Evaluation of Combined Sensitising and Hypomethylating Therapy Outcomes in AML PDX
Brief Title: Evaluation of Combined Sensitising and Hypomethylating Therapy Outcomes in AML PDX
Acronym: COSMOS-Avatar
Status: Recruiting | Type: Observational
Sponsor: Clinical Hub for Interventional Research (CHOIR) (Other Government)
Collaborators: Cancer Institute NSW (Unknown); The University of New South Wales (Other); Australian National University (Other)
Responsible Party: Sponsor
Other Study IDs: 24-M-003
Record Dates: First submitted 2025-01-09; First posted 2025-01-20 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-06

CONDITIONS: AML - Acute Myeloid Leukemia
Keywords: AML; Acute Myeloid Leukemia; PDX; Patient-derived xenografts
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Peripheral blood and bone marrow aspirate research samples will be collected. After research samples have been processed, analysed, and stored for study endpoint evaluation, as specified in this protocol, the remaining specimens will be stored indefinitely for use in future related research.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Cohort 1: Individuals diagnosed with or suspected of acute myeloid leukemia (AML) who are not planned for intensive chemotherapy and are commencing venetoclax + azacitidine therapy.
- Cohort 2: Individuals who have relapsed following, or are refractory to, intensive chemotherapy or hematopoietic stem cell transplantation, commencing venetoclax + azacitidine therapy.

SUMMARY:
The goal of this observational study is to develop new ways to test new drug combinations to kill tumour cells, in patients with acute myeloid leukemia (AML). The main questions it aims to answer are:

* Are there new ways to speed up discovery of better treatments for AML patients using AML cells from individual from patients in special mice that can accept human tissue?
* Do these mice show treatment responses that are similar to the individual AML patient from whom cells were derived?

Participants with AML who are taking standard of care treatment of venetoclax and azacitidine will be asked to donate blood and bone marrow samples for this study.

DETAILED DESCRIPTION:
Treatment options for patients with acute myeloid leukemia (AML) who are unfit or refractory to intensive chemotherapy, or who have relapsed after hematopoietic stem cell transplantation, remain limited. Hypomethylating agents (HMAs) are effective in prolonging patient survival, but they are often associated with adverse events and their therapeutic effects are temporary. By elucidating the resistance mechanisms used by AML cells, we have identified drugs that selectively sensitise these tumour cells to HMAs, with minimal toxicity to healthy blood cells. Patient-derived xenografts (PDX) have emerged as a valuable tool for drug testing in cancer research. They can better replicate the primary tumour and its environment in vivo, mimicking the disease progression and treatment responses of their corresponding donor with superior fidelity and predictive potential compared to current in vitro systems. The COSMOS-Avatar study aims to establish a drug testing platform to guide precision therapies tailored to defined tumour profiles. Tumour cells obtained over two years through altruistic donation for research will be used to generate AML PDX mouse models or avatars that will be used to compare standard of care and multiple candidate therapies simultaneously. Promising drug combinations identified through the COSMOS-Avatar study will proceed to a dedicated independent Phase I clinical trial platform to accelerate drug discovery and development of AML therapies.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18 years and above
2. Patients with suspicion of AML requiring screening procedures
3. Documented diagnosis of AML by WHO Classification and/or International Consensus Classification.

   * Regardless of the number and type of prior lines of therapy or eligibility for allogeneic stem cell transplantation.
   * All AML subtypes are eligible.
   * Concurrent participation in clinical trials is allowed.
4. Documented myeloblast percentage ≥20% in the bone marrow or peripheral blood within 12 weeks of C1D1 confirmed by bone marrow aspirate or peripheral blood smear.
5. Planned to commence venetoclax and azacitidine therapy.
6. Provision of written informed consent prior to any study-related assessments or procedures being carried out.

Exclusion Criteria:

1. Presence of any condition that, by assessment of the Investigator, would compromise the safety of the patient if they participated, the quality of trial data, or their adherence to the study-specified procedures.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Study population is people who have recently been diagnosed with or are suspected of having AML and undergoing investigational procedures, and whose doctor plans to start them on venetoclax and azacitidine. Around 25 people from different hospitals in Australia will take part in this project.
Sampling Method: Non-Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2028-02 (Estimated); Study Completion 2030-03 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint - Generation of ≥20 adult AML PDX models with clinically annotated samples, including treatment regimen and clinical outcome | From enrolment (i.e., C1D1 of Ven+AZA treatment) up to end of treatment or 52 weeks post C1D1 (whichever applies first)
  The outcome measures are 1) establish an adult AML PDX drug testing platform; 2) determine how accurately the AML PDX model replicates the clonal architecture and cellular characteristics of the original tumour by comparing donors' samples to AML PDX samples; 3) compare efficacy of standard of care and candidate therapies by engrafting multiple immune-deficient mice with the same donor sample; and 4) biomarker discovery through correlation of treatment response and single-cell and cytokine analysis.

SECONDARY OUTCOMES:
Secondary Endpoint - Frequency and phenotype of leukemic cells measured by flow cytometry in AML PDX models and primary donor samples before and after VEN+AZA treatment. | From enrolment (i.e., C1D1 of Ven+AZA treatment) up to end of treatment or 52 weeks post C1D1 (whichever applies first)
  A) Peripheral blood and bone marrow samples will be collected from Cohort 1 and Cohort 2 participants at baseline and relapse and will undergo molecular and cellular characterisation, these samples will be used to generate AML PDX models. B) Cells isolated from participant samples will be used to generate adult AML PDX models by reconstituting immune-deficient mice and expand the cell stock in vivo. Expanded cells will be used to reconstitute additional immune-deficient mice. C) Samples will be collected from immune-deficient mice before and after treatment to assess the efficacy of individual treatments. Participant and PDX samples will also be compared to assess the fidelity of the PDX model to their matching donor.

CONTACTS AND LOCATIONS:
Overall Officials: John Pimanda, Professor, Principal Investigator — University of New South Wales
Locations (4):
- Australia (4):
  - Canberra Health Services, Canberra, Australian Capital Territory
  - Prince of Wales Hospital, Sydney, New South Wales
  - Royal North Shore Hospital, Sydney, New South Wales
  - Westmead Hospital, Westmead, New South Wales

IPD SHARING:
Plan to Share IPD: No